CLINICAL TRIAL: NCT00002069
Title: A Study of DTC in Patients With AIDS and AIDS Related Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merieux Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 010A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-07

CONDITIONS: HIV Infections
Keywords: Ditiocarb; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ditiocarb

INTERVENTIONS:
Drug: Ditiocarb sodium

SUMMARY:
To determine if ditiocarb sodium (sodium diethyldithiocarbamate; DTC) restores immune and host defense function; if DTC ameliorates the AIDS related complex (ARC) symptoms in patients with AIDS and ARC; if DTC prevents progression from ARC to AIDS or progression of AIDS; and if DTC prolongs survival in AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Active opportunistic infection or progressive Kaposi's sarcoma (KS).
* Dementia.
* Lymphoma.

Concurrent Medication:

Excluded within 3 weeks of study entry:

* Other experimental AIDS therapy.

Patients with the following are excluded:

* Active opportunistic infection or progressive Kaposi's sarcoma (KS).

Patients must be either HIV seropositive or have AIDS or AIDS related complex (ARC) and have life expectancy of at least 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Univ of Arizona / Arizona Cancer Ctr, Tucson, Arizona
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Portion Med Group, Sherman Oaks, California
  - Florida Keys Memorial Hosp, Key West, Florida
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Dr Gary Brewton, Houston, Texas

REFERENCES:
- [Background] Hersh EM, et al. A randomized, double-blind, placebo-controlled trial of diethyldithiocarbamate (Ditiocarb, Imuthiol(R) in patients with ARC and AIDS. Int Conf AIDS. 1990 Jun 20-23;6(3):208 (abstract no SB489)